CLINICAL TRIAL: NCT00968058
Title: Temporal Variation of the Leak Pressure of Uncuffed Pediatric Endotracheal Tubes Following Intubation: A Prospective Observational Study
Brief Title: Leak Pressure of Uncuffed Pediatric Endotracheal Tubes
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kirk Lalwani, Associate professor Anesthesiology and Pediatrics, Oregon Health and Science University
Other Study IDs: IRB00005347
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Intubation, Endotracheal; Leak Pressure
Keywords: Leak Pressure; Intubation, Endotracheal; Pediatric; Temporal Variation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Leak Test Recording — Recording of the Leak Pressure by the Leak Test at 0, 5, 10, 15, 20, 30 min timepoints

SUMMARY:
Children and adults frequently need a 'breathing tube' when having anesthesia for surgery. The breathing tube is usually inserted after the anesthesia doctor puts a patient to sleep with medicine, so they do not feel the breathing tube. In children, there is often a leak of air between the tube and the windpipe, as the tube is not an exact fit. Anesthesia doctors usually listen for this leak around the tube by listening to the chest with a stethoscope while gently filling the lungs with oxygen from the anesthesia machine. The leak tells them if the tube is the correct size, or too small, or too tight. If it is too small, or too tight, they usually change the tube for a better fit.

The purpose of this study is to see what happens to this leak in the 30 minutes after the tube is placed. No one really knows if the leak gets bigger, smaller, or stays the same. Knowing what happens to the leak will help anesthesia doctors to decide whether to change the breathing tube or not. This is important, as a tube that is too tight can lead to breathing difficulty after removing the tube at the end of surgery, and a tube that is too small may make it difficult for the breathing machine to work effectively for the patient as a result of a large leak of air or oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-7 years of age
* Surgery with planned endotracheal intubation using an uncuffed ETT.
* ASA 1-3
* Supine position

Exclusion Criteria:

* Lack of parental consent
* Rapid sequence induction with cricoid pressure
* Use of neuromuscular blocking agent/s for intubation.
* Active gastroesophageal reflux disease
* Active upper respiratory tract infection
* Chronic active lung disease requiring frequent treatment such as asthma, or chronic lung disease of prematurity etc.
* Surgery in the lateral or prone position
* Oropharyngeal, neck , laryngeal, or laparoscopic surgery
* Tracheostomy in-situ
* History of previous laryngeal or tracheal surgery
* History of tracheal or laryngeal abnormalities, or stridor of unknown origin.
* History of symptomatic neuromuscular disease or paralysis
* History or features suggestive of a difficult airway on pre-anesthetic evaluation and physical examination.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing surgical procedures at Oregon Health & Science University
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in leak pressure following endotracheal tube placement | Thirty minutes after tube placement

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Lalwani, MD, Principal Investigator — Oregon Health and Science University; Shreya J Patel, BS, Study Director — University of Arizona College of Medicine; Jeffrey Koh, MD, Study Director — Oregon Health and Science University; Rochelle Fu, PhD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States